CLINICAL TRIAL: NCT07224087
Title: Development of a Multiple Health Behavior Change Intervention for Weight Loss and Smoking Cessation for Pre-Bariatric Surgery Patients
Brief Title: Development of a MHBC Intervention for Weight Loss and Smoking Cessation for Pre-Bariatric Surgery Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Society for Metabolic and Bariatric Surgery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000041069
Record Dates: First submitted 2025-10-23; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Smoking Cessation; Bariatric Surgery Patients
MeSH Terms: conditions — Obesity; Smoking Cessation | interventions — Naltrexone; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: All participants will receive the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Participants will receive the multiple health behavior change intervention with combined medication (Naltrexone 50mg/day; Bupropion Extended Release 300mg/day) and behavior therapy (Cognitive-Behavioral Therapy) for 4 months.
  Interventions: Drug: Naltrexone Hydrochloride; Drug: Bupropion HCl Extended Release; Behavioral: Cognitive-Behavioral Therapy

INTERVENTIONS:
Drug: Naltrexone Hydrochloride — Participants will be given 50mg/day of Naltrexone for 4 months.
Drug: Bupropion HCl Extended Release — Participants will be given 300mg/day of Bupropion for 4 months. Bupropion will be taken twice daily (150mg in the morning, followed by 150mg in the late afternoon/early evening).
Behavioral: Cognitive-Behavioral Therapy — Participants will receive cognitive-behavioral therapy for weight loss and smoking cessation. Participants will meet with their assigned study clinician weekly for 60 minutes for 4 months.

SUMMARY:
The purpose of this research study is to develop and pilot a multiple health behavior change intervention for weight loss and smoking cessation using medication (Naltrexone + Bupropion) and behavior therapy in adults seeking bariatric surgery.

DETAILED DESCRIPTION:
Smoking prevalence among pre-bariatric surgery patients is estimated to be as high as 40%. In addition to quitting smoking, patients are expected to lose weight before surgery, which is challenging as smoking cessation is associated with weight gain. Pre-bariatric surgery patients would significantly benefit from a tailored multiple health behavior change intervention targeting weight loss and smoking cessation concurrently, yet no such interventions have been examined within this patient population.

This study aims to develop and pilot a multiple health behavior change intervention with combined behavioral and pharmacotherapy (Naltrexone + Bupropion) for weight loss and smoking cessation for adults seeking bariatric surgery. This pilot will evaluate the feasibility and acceptability of the intervention, as well as use a mixed methods approach for intervention refinement. Weight loss and smoking cessation will be assessed post-treatment. This study will provide important preliminary data needed to develop an effective intervention that will address weight loss and smoking cessation concurrently, which is needed to improve bariatric surgery utilization and reduce risk for smoking relapse post-surgery for this high-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* Be actively considering bariatric surgery.
* Smoke at least 5 cigarettes daily for the past 3 months.
* Have a BMI ≥ 30.0 kg/m2.
* Not currently taking medications that interact with Naltrexone or Bupropion (e.g., opiates, benzodiazepines).
* No history of medical conditions that are contraindicated with Naltrexone or Bupropion (e.g., seizure disorders, uncontrolled hypertension, cardiac issues including history of heart attacks, heart disease, or stroke, history of anorexia or bulimia nervosa).
* Physically well enough to participate in the intervention (e.g., able to walk independently).
* Speak/read/write in English.
* Be 18-65 years old.
* Not currently pregnant or breastfeeding or have plans to become pregnant or breastfeed during the study.
* No active suicidal or homicidal ideation.

Exclusion Criteria:

* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently taking a medication that is contraindicated to Naltrexone or Bupropion (e.g., MAOIs, opiates).
* Has a history of allergy or sensitivity to Naltrexone or Bupropion.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression).
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute.
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled Type I or Type 2 diabetes mellitus.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary, or gallbladder disease, or any other unstable medical disorder.
* Is breast-feeding or is pregnant or is not using a reliable form of birth control.
* Reports active suicidal or homicidal ideation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Study enrollment to assess Feasibility | 16 weeks
  Number of participants enrolled out of participants screened
Mean number treatment sessions attended to assess Feasibility | 16 weeks
  Mean number of treatment sessions attended
Retention to assess Feasibility | 16 weeks
  Retention will be measured as the percent of participants that attend the post treatment assessment
Treatment credibility and satisfaction to assess Acceptability | 16 weeks
  Treatment credibility and satisfaction will be assessed via self-report at post-treatment. Acceptability measured as the percent of participants that agree the intervention is acceptable.
Percent weight change | Baseline and Week 16
  Percent weight change will be calculated from baseline to post-treatment.
Smoking cessation, as measured by exhaled carbon monoxide | Baseline, Week 4, Week 8, Week 12, Week 16
  Smoking cessation will be evaluated biochemically, through mean exhaled carbon monoxide concentration.
Smoking cessation, as measured by timeline followback interview | Baseline, Week 4, Week 8, Week 12, Week 16
  Smoking cessation will be evaluated behaviorally, through point prevalence abstinence data obtained by timeline followback interviews.

SECONDARY OUTCOMES:
Nicotine dependence, as measured by the Fagerstrom Test for Nicotine Dependence | Baseline and Week 16
  The Fagerstrom Test for Nicotine Dependence is a self-report measure that classifies level of nicotine dependence. Participants respond to a series of questions assessing time of first cigarette after waking, difficulty refraining from smoking in places where smoking is prohibited, and frequency of smoking. Total score range 0-10 with higher scores indication more nicotine dependence.
Depressive symptomatology, as measured by the Patient Health Questionnaire-9 | Baseline and Week 16
  The Patient Health Questionnaire-9 is a brief, psychometrically sound, and widely used self-report measure of depression in diverse medical settings. The total score on the PHQ-9 ranges from 0 to 27, with higher scores indicating greater severity of depressive symptoms.
Physical activity, as measured by the Global Physical Activity Questionnaire (GPAQ) | Baseline and Week 16
  GPAQ is a validated self-report assessment of physical activity and sedentary behavior. GPAQ does not have a single fixed total score range but a score is calcualed in METs-minutes per day. Participants are classified as "active" if they meet or exceed 600 METs-minutes per week.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Smith, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chow A, Neville A, Kolozsvari N. Smoking in bariatric surgery: a systematic review. Surg Endosc. 2021 Jun;35(6):3047-3066. doi: 10.1007/s00464-020-07669-3. Epub 2020 Jun 10. PMID 32524412